CLINICAL TRIAL: NCT00020696
Title: A Phase II Evaluation of Tirapazamine (NSC #130181, IND #46,525) in Combination With Cisplatin in Recurrent Platinum Sensitive Ovarian or Primary Peritoneal Cancer
Brief Title: Tirapazamine Plus Cisplatin in Treating Patients With Persistent or Recurrent Ovarian Epithelial or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068705; GOG-0146M
Record Dates: First submitted 2001-07-11; First posted 2004-02-04 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2008-03

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Cisplatin; Tirapazamine

INTERVENTIONS:
Drug: cisplatin
Drug: tirapazamine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining tirapazamine with cisplatin in treating patients who have recurrent ovarian epithelial or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of tirapazamine and cisplatin in patients with persistent or recurrent platinum-sensitive ovarian epithelial or primary peritoneal carcinoma.
* Determine the nature and degree of toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive tirapazamine IV over 2 hours followed 1 hour later by cisplatin IV over 30 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 20-65 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed persistent or recurrent ovarian epithelial or primary peritoneal carcinoma
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* Platinum-sensitive disease

  * Treatment-free interval of more than 6 months without clinical evidence of progressive disease after a response to a platinum compound
* One prior chemotherapy regimen containing cisplatin or another platinum compound for primary disease required

  * Initial treatment may include high-dose therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment
  * Patients not previously treated with paclitaxel may receive a second regimen containing paclitaxel
  * No additional cytotoxic chemotherapy (including retreatment with initial regimens) for recurrent or persistent disease
* Ineligible for a higher priority GOG protocol (any active GOG phase III protocol for the same patient population)

  * Treatment-free interval of more than 12 months if non-platinum-based GOG-0146 series protocol is active concurrently with this protocol

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No prior or concurrent myocardial infarction or ischemic heart disease

Other:

* No active infection requiring antibiotics
* No sensory or motor neuropathy greater than grade 1
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic or immunological agents directed at malignant tumor

Chemotherapy:

* See Disease Characteristics
* Recovered from prior chemotherapy
* No prior tirapazamine

Endocrine therapy:

* At least 1 week since prior hormonal therapy directed at malignant tumor
* Concurrent hormone replacement therapy allowed

Radiotherapy:

* Recovered from prior radiotherapy
* No prior radiotherapy to site(s) of measurable disease used on this study
* No prior radiotherapy to more than 25% of bone marrow

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* No prior cancer treatment that would preclude study
* At least 3 weeks since other prior therapy directed at malignant tumor

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Covens, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (54):
- United States (50):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Australia New Zealand Gynaecological Oncology Trials Group, Camperdown, New South Wales, Australia
- Canada (2):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
- University of Birmingham, Birmingham, England, United Kingdom

REFERENCES:
- [Result] Covens A, Blessing J, Bender D, Mannel R, Morgan M; Gynecologic Oncology Group. A phase II evaluation of tirapazamine plus cisplatin in the treatment of recurrent platinum-sensitive ovarian or primary peritoneal cancer: a Gynecologic Oncology Group study. Gynecol Oncol. 2006 Mar;100(3):586-90. doi: 10.1016/j.ygyno.2005.09.032. Epub 2005 Oct 24. PMID 16249022